CLINICAL TRIAL: NCT03034707
Title: Interference of Biotin Supplementation in Biotin-streptavidin Platforms for Hormone Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Johns Hopkins University (Other); Boston Medical Center (Other); Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1602M84022
Record Dates: First submitted 2017-01-17; First posted 2017-01-27 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Thoracic Diseases; Parathyroid Diseases
Keywords: biotin pharmacokinetic; biotinylated assay; hormone measurement; thyroid; parathyroid; prolactin
MeSH Terms: conditions — Thoracic Diseases; Parathyroid Diseases; Thyroid Diseases | interventions — Biotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biotin arm (Experimental): biotin 10 mg/day for 7 days
  Interventions: Dietary Supplement: biotin

INTERVENTIONS:
Dietary Supplement: biotin

SUMMARY:
The B vitamin biotin is widely available as an over the counter supplement, often advertised and used to promote health of hair, skin and nails. Commercially available over the counter biotin supplements contain dose ranges up to 10 mg/day (ie 333 times higher than the recommended dietary allowance). The biotin molecule is also sometimes used as part of the lab technology to measure hormone and protein levels in the blood. It is possible that high doses of ingested biotin may interfere with accurate hormone or protein measurement using biotin related in vitro measurement systems. Such interference, if present, could lead to misdiagnosis. The study will analyze laboratory levels obtained with streptavidin-biotin assay systems while ingesting biotin in currently available high dose supplements. The data will be compared to measurements obtained prior to and one week after stopping the biotin supplement.

DETAILED DESCRIPTION:
Specimens will be collected by venipuncture at 3 time points, including baseline (time 0), after one week of biotin supplementation (time 1, day 7), and then one week later (time 2, day 14). The time 1 specimen will be drawn approximately 2 hours after the last ingested dose of biotin on day 7. Specimen collection will include three 10 ml red top (no gel) tubes at each timepoint.

Specimens will be separated for isolation of serum using routine methods of the clinical chemistry laboratory. Serum will be stored at -80 degrees C until batch measurements as described Measurements Biotin levels will be measured on each sample. Hormone measurements will be performed using specific commercially available streptavidin-biotin assays and using different analyzers as indicated below. Immunoassay methods, not employing biotin-streptavidin methodology, will be used for negative assay controls.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults

Exclusion Criteria:

1. Pregnancy or lactation
2. Known thyroid disease (goiter, abnormal thyroid state),
3. Thyroid hormone treatment,
4. Over the counter dietary/ nutritional supplement use currently or within the last 2 weeks (excluding standard multivitamin preparations containing no more than 100% of the daily value for biotin and calcium),
5. Anticonvulsants,
6. Night shift work, smokers, adults lacking capacity to consent for themselves

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Hormone measurements TSH, PTH, Total T4, free T4, total T3, free T3, prolactin | Change from baseline, at 7 days, at 14 days
  Hormone measurements using biotinylated assay conducted in certified labratory using the standard lab ranges for each test.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn A Burmeister, MD, Principal Investigator — Univ of Minnesota; Angela Radulescu, MD, Study Director — Univ of Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiume MZ; Cosmetic Ingredient Review Expert Panel. Final report on the safety assessment of biotin. Int J Toxicol. 2001;20 Suppl 4:1-12. PMID 11800048
- [Background] Meany DL, Jan de Beur SM, Bill MJ, Sokoll LJ. A case of renal osteodystrophy with unexpected serum intact parathyroid hormone concentrations. Clin Chem. 2009 Sep;55(9):1737-9. doi: 10.1373/clinchem.2008.121921. No abstract available. PMID 19717659
- [Background] Kwok JS, Chan IH, Chan MH. Biotin interference on TSH and free thyroid hormone measurement. Pathology. 2012 Apr;44(3):278-80. doi: 10.1097/PAT.0b013e3283514002. No abstract available. PMID 22437752
- [Background] Wijeratne NG, Doery JC, Lu ZX. Positive and negative interference in immunoassays following biotin ingestion: a pharmacokinetic study. Pathology. 2012 Dec;44(7):674-5. doi: 10.1097/PAT.0b013e32835a3c17. No abstract available. PMID 23089740
- [Derived] Li D, Radulescu A, Shrestha RT, Root M, Karger AB, Killeen AA, Hodges JS, Fan SL, Ferguson A, Garg U, Sokoll LJ, Burmeister LA. Association of Biotin Ingestion With Performance of Hormone and Nonhormone Assays in Healthy Adults. JAMA. 2017 Sep 26;318(12):1150-1160. doi: 10.1001/jama.2017.13705. PMID 28973622